CLINICAL TRIAL: NCT01250899
Title: Vitamin D, Immune Activation, and Metabolic Abnormalities in HIV-Infected Patients on Antiretroviral Therapy
Brief Title: Vitamin D in HIV-Infected Patients on HAART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jordan E. Lake M.D., M.D., University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARE Vitamin D
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Vitamin D Deficiency; HIV
Keywords: HIV; Vitamin D; HAART
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D Sufficient (No Intervention): HIV-infected men and women with HIV-1 viral load <200 copies/mL on stable ART and 25(OH)D level ≥30ng/mL receive no intervention.
- Vitamin D Insufficient (Experimental): HIV-infected men and women with HIV-1 viral load <200 copies /mL on stable ART and 25(OH)D level <30ng/mL receive 50,000 IU twice weekly for 5 weeks followed by 2000 IU daily to complete 12 weeks.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 50,000 IU vitamin D3 twice weekly for 5 weeks, followed by 2000 IU daily maintenance supplementation to complete 12 weeks. At the end of the 12-week period, 25(OH)D levels will be checked. If the subject is still deficient, he/she may undergo a second period of supplementation (at the discretion of their provider) to complete a total of 24 weeks. After 24 weeks, we anticipate all subjects will be kept on daily maintenance supplementation by their primary physicians.
  Arms: Vitamin D Insufficient

SUMMARY:
This is a research study to look at vitamin D deficiency (low levels) in men and women with HIV. As part of your regular medical care, you will be screened for vitamin D deficiency. If your levels are low, and you choose to start using vitamin D supplements, the investigators would like to take some blood before and after you start using vitamin D to see how this affects your levels of HIV, T cells, cholesterol, and other blood levels. The investigators will provide you with vitamin D supplements for the first 24 weeks (6 months) of the study. If you and your physician decide that you should continue taking vitamin D supplements after that time, you will be responsible for purchasing your own vitamin D supplements.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive men and women age 18 and older.
* HIV-1 RNA documented to be < 200 copies/mL on their current ART regimen, with supporting viral load documentation in the 24 weeks prior to study entry.
* Subjects must receive primary HIV care at the UCLA CARE center.
* Subjects must be undergoing screening for vitamin D deficiency by their primary care provider at the time of study entry, or have undergone vitamin D screening in the 90 days prior to consent without yet initiating vitamin D supplementation (for insufficient subjects).
* Ability and willingness of subject to provide informed consent

Exclusion Criteria:

* Use of vitamin D supplementation (not including 400 IU daily, the amount in a standard multivitamin) at the time of screening.
* HIV-infected subjects not on ART.
* HIV-infected subjects not suppressed on their current ART regimen (HIV-1 RNA > 200 copies/mL in the 6 months prior to screening).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Currier, M.D., Study Director — University of California, Los Angeles; Jordan Lake, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA CARE Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D Sufficient: HIV-infected men and women on stable ART underwent routine serum 25(OH)D screening. Persons with HIV-1 RNA <200 copies/mL and reported taking daily vitamin D <400 IU were eligible to participate. Subjects with 25(OH)D ≥30ng/mL had a baseline visit only, and did not receive vitamin D supplementation.
- Vitamin D Insufficient: HIV-infected men and women on stable ART underwent routine serum 25(OH)D screening. Persons with HIV-1 RNA <200 copies/mL and reported taking daily vitamin D <400 IU were eligible to participate. Subjects with 25(OH)D <30ng/mL received open-label, oral vitamin D3 50,000 IU twice weekly for 5 weeks, then 2000 IU daily to complete 12 weeks. Serum 25(OH)D levels were measured at baseline, 12 weeks and 24 weeks.
Period: Overall Study
Arm/Group | Vitamin D Sufficient | Vitamin D Insufficient
Started | 40 | 82
Completed | 40 | 82
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: HIV-infected men and women with HIV-1 RNA <200 copies/mL on stable ART and daily vitamin D <400IU were enrolled
Groups:
- Vitamin D Sufficient: HIV-infected men and women on stable ART with HIV-1 RNA <200 copies/mL and reported taking daily vitamin D <400 IU were eligible to participate. Subjects with 25(OH)D ≥30ng/mL had a baseline visit only, and did not receive vitamin D supplementation.
- Vitamin D Insufficient: HIV-infected men and women on stable ART with HIV-1 RNA <200 copies/mL and reported taking daily vitamin D <400 IU were eligible to participate. Subjects with 25(OH)D <30ng/mL received open-label, oral vitamin D3 50,000 IU twice weekly for 5 weeks, then 2000 IU daily to complete 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Vitamin D Sufficient | Vitamin D Insufficient | Total
Number analyzed (Participants) | 40 | 82 | 122
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [43 to 56] | 48 [39 to 57] | 48 [39 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 38 | 78 | 116

OUTCOME MEASURES:

1. Primary Outcome: Success Rate in Achieving a 25(OH)D Level ≥30ng/mL After 12 Weeks of Oral Vitamin D Supplementation.
Description: Percentage of participants successfully repleted to 25(OH)D ≥30ng/mL after 12 weeks of oral vitamin D supplementation.
Time Frame: 12 weeks
Population: After 12 weeks of oral vitamin D supplementation, serum 25(OH)D levels were measured in the Vitamin D Insufficient arm. 81% (n=66) of insufficient persons achieved 25(OH)D ≥30ng/mL (p=0.32 vs. historical controls).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Vitamin D Insufficient: Baseline 25(OH)D <30 ng/mL received 12 weeks of oral vitamin D supplementation. Serum 25(OH)D levels were measured at baseline, 12 weeks and 24 weeks.
Arm/Group | Vitamin D Insufficient
Number analyzed (Participants) | 82
percentage of participants | 81 [70 to 88]
Statistical Analysis 1: Comparison: Vitamin D Insufficient; We predicted that HIV-infected subjects would have a 70% twelve-week repletion success rate compared to 85% among historical controls.Eighty subjects provided 91% power to detect a 12-week repletion rate statistically different than 85% (95% confidence interval (CI) 60%, 80%); Test type: Superiority or Other; p < 0.05, Exact binomial; Percentage of 12-wk 25(OH)D ≥30ng/mL = 70, 95% CI 2-sided [60 to 80] — The primary endpoint (mean change in 25(OH)D following 12 weeks of vitamin D repletion in vitamin D insufficient subjects) was dichotomized to success or failure to achieve a week twelve 25(OH)D level ≥30ng/mL

ADVERSE EVENTS:
Time Frame: 12 weeks, 24 weeks
Groups:
- Vitamin D Insufficient: 25(OH)D <30 mg/mL at study entry (i.e. group of patients receiving vitamin D supplementation).
Arm/Group | Vitamin D Insufficient
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

LIMITATIONS AND CAVEATS:
This trial was prospective, but open label and not randomized. However, randomization to placebo would not have been clinically appropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No